CLINICAL TRIAL: NCT01899664
Title: Study of the Surgical Treatment of Cervical Spinal Cord Injuries With Nerve Transfers to Restore Upper Extremity and Hand Function
Brief Title: Upper Extremity Surgery in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201205104
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Quadriplegia; Spinal Cord Diseases; Spinal Cord Injuries
Keywords: peripheral nerves; quadriplegia; nerve transfer; surgical procedures, operative; hand; upper extremity; quality of life
MeSH Terms: conditions — Quadriplegia; Spinal Cord Diseases; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Subjects will undergo the following:
  A full International Standards for Neurological Classification of SCI exam will be completed to determine exact function and type of spinal cord injury.
  A phone interview will be completed at both preoperative and postoperative time points.
  Quality of life before and after surgical intervention will be derived from standardized questionnaires: Spinal Cord Independence Measure (SCIM), SF-36, Novak scale, and pain questionnaires.
  Additional qualitative and quantitative data on donor and recipient nerve function and tissue will be derived from preoperative electrodiagnostic studies.
  Specimens of the donor and recipient nerve are collected for histologic analysis during the operative procedure. Those trimmed nerve specimens are then analyzed for clinical purposes to give patients an idea of expected outcome in a more timely fashion.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary Study Population (Other): Study participants (primary study population) will include patients with spinal cord injury at the mid cervical level who are undergoing evaluation for possible surgical treatment with nerve transfers and or tendon transfer/tenodesis to improve their upper extremity function. All enrolled participants will receive the same standard of care surgical procedures.
  Interventions: Procedure: Nerve Transfer Surgery

INTERVENTIONS:
Procedure: Nerve Transfer Surgery — Unilateral surgery will be performed under general non-paralytic anesthesia and no-tourniquet conditions to allow for responsive nerve simulation.

SUMMARY:
The goal of the investigators work is to establish how nerve transfers can be best used to improve upper extremity function in patients with cervical level spinal cord injury (SCI). The investigators' hypothesis is that nerve transfers are safe and effective and will improve function and quality of life in patients with loss of upper function due to spinal cord injury. The investigators plan on looking at upper limb function, and health-related quality of life in patients before and after surgery to better understand how patients benefit from these treatments.

A nerve transfer procedure can be used to rewire the system to make some muscles work again following SCI. The nerve transfer procedure (which is done in the arm and not at the level of the spinal cord) can be used to bypass the damaged area and to deliver a signal from the brain to a muscle that became disconnected following that injury. A donor nerve is taken from another muscle whose use is not essential and then transferred to help in providing more a more critical function.

For example, one type of nerve transfer is done to restore the lost ability to pinch or grasp small objects between the fingers that occurs in many patients with cervical SCI. In this surgery, a donor nerve that normally helps flex the elbow. This nerve can be used because the biceps muscle is also working to flex the elbow. This donor nerve is cut and re-attached to the nerve going to muscles in the forearm that provide pinch by bending the tips of the thumb and index finger.

Because the nerve transfer procedure involves cutting and reattaching nerve and muscle tissues, time is required to regenerate working connections between the nerves and muscle as well as to allow the brain to relearn how to use and strengthen that muscle.

DETAILED DESCRIPTION:
Background/Readiness

Cervical spinal cord injury (SCI) is a life altering injury that results in profound loss of upper limb function. Nerve transfer surgery has transformed the field of peripheral nerve injury surgery, allowing remarkable restoration of upper limb motor function. The investigators expanded use of nerve transfer surgery to cervical SCI patients and are the first center to successfully restore volitional hand function in a patient with a C7 motor level injury (now 3 years post-surgery). Results in 7 more patients show early functional gains at 3-6 months post-surgery (most gains are expected at 12 months and these patients are still early in their course). The proposed study will obtain formative outcomes data from a pilot investigation of nerve transfer surgery to restore upper extremity function in patients with cervical SCI.

Upper extremity and hand function is essential to basic activities of daily living and independence; patients with cervical SCI rate this as more important than walking and sexual performance. Restoration of critical upper extremity and hand function requires the unique expertise and technical skill of hand surgeons; traditionally tendon transfer/tenodesis are used. Although studies report reasonable outcomes in SCI patients for this procedure, use is limited particularly in the US.

Nerve transfers offer an alternative and promising approach. In peripheral nerve injury, nerve transfers are well-established, safe and are often the treatment of choice. A nerve transfer uses an expendable donor nerve and coapts this to a nonfunctional recipient nerve to restore volitional motor function. Since a nerve transfer reinnervates the musculotendinous unit responsible for the absent but desired function, this procedure: 1) does not have the biomechanical limitations of tendon transfers; 2) can use expendable donor nerves whose muscles cannot be used for tendon transfer (i.e. the brachialis); and 3) a single donor nerve can provide more than one function via reinnervation of multiple muscles. Most importantly for SCI patient acceptability, nerve transfers do not require prolonged periods of immobilization; early resumption of activity is encouraged.

Preliminary Data:

Case reports offer early evidence that this novel application of nerve transfers may be a better alternative to tendon transfers in SCI. Based on our extensive experience with nerve transfers in peripheral nerve injury, we expect this approach will have a profound impact on improving function, independence and health-related quality of life (QoL).

The purpose of this study is to provide evidence on the feasibility, safety, and outcomes of nerve transfers in SCI patients via systematically collected data and to evaluate patients' perspective of the benefits and disadvantages of nerve transfers. These data are vital for patient selection, patient and surgeon education, and adaptation of this well-established technique to this unique and traditionally underserved patient population.

Hypothesis and Approach:

Hypothesis: Nerve transfers are safe, effective procedures that have a role in the treatment armamentarium of cervical SCI associated upper extremity dysfunction.

Aim 1: To document the safety, time course and improvement (potential for nerve transfers to improve functional outcomes) by assessing pre and post-operative function.

Aim 2: To evaluate the feasibility and suitability of nerve transfers through multidisciplinary evaluation, electrodiagnostic testing, ultrasound, and nerve specimen examination and correlation with the clinical outcome.

Aim 3: To assess patient satisfaction with and acceptability for this treatment by use of semi-structured patient interviews.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cervical level spinal cord injury
* some upper extremity dysfunction (ex: lack of wrist extension or hand function)
* greater then 6 months post-injury or with stable neurologic function for at least 6 months post-injury
* good access to and ability to pay for hand and physical therapy
* ability to comply and participate in rigorous post-surgical therapy regimen

Exclusion Criteria:

* severe autonomic dysreflexia
* open pressure sores or other wounds
* respiratory insufficiency
* untreated urinary tract infections
* lack of access to physical therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Upper extremity function. | change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  Upper extremity function as measured by manual muscle testing and range of motion as well as the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) test (this is a standardized functional test to assess upper extremity function in patients with spinal cord injury) and International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) test (this is an examination used to determine the motor and sensory impairment and severity of a spinal cord injury).

SECONDARY OUTCOMES:
Health related quality of life. | change from baseline at 6, 12, 24, 30 and 36 months post-surgery
  The Short Form (SF) -36, Spinal Cord Independence Measure (SCIM), Canadian Occupational Performance Measure (COPM) will be used to provide information about the patients quality of life and function.
  Semi-structured interviews will be performed at 12-18 months following surgery to gain information about patient satisfaction, acceptability, and the subjective experience of the surgical intervention, therapy and functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ida K. Fox, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Division of Plastic Surgery, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Nerve Transfers to Restore Upper Extremity Function in Cervical Spinal Cord Injury: Update and Preliminary Outcomes. Plast Reconstr Surg. 2015 Oct;136(4):780-792. doi: 10.1097/PRS.0000000000001641. PMID 26397252
- [Result] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Use of peripheral nerve transfers in tetraplegia: evaluation of feasibility and morbidity. Hand (N Y). 2015 Mar;10(1):60-7. doi: 10.1007/s11552-014-9677-z. PMID 25767422
- [Derived] Hill EJR, Fox IK. Current Best Peripheral Nerve Transfers for Spinal Cord Injury. Plast Reconstr Surg. 2019 Jan;143(1):184e-198e. doi: 10.1097/PRS.0000000000005173. PMID 30589809
- See also: Patient information and intake forms. — http://nerve.wustl.edu/nd_C6-C7_spinal_injury.php